CLINICAL TRIAL: NCT07113691
Title: Iadademstat and Radiation Therapy With Atezolizumab in Extensive Stage Small-cell Lung Cancer (ES-SCLC) Patients With Persistent, Recurrent or Progressive Disease After First Line Systemic Therapy
Brief Title: Iadademstat + SBRT With Atezo in ES-SCLC
Acronym: TIARA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry); Oryzon Genomics S.A. (Industry)
Responsible Party: Principal Investigator, Anne Chiang, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000039106
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Keywords: persistent, recurrent or progressive disease after first line systemic therapy
MeSH Terms: conditions — Recurrence | interventions — iadademstat; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Iadademstat + Atezolizumab (Experimental): The first three participants will start iadademstat at a dose of 600ug PO weekly (DL 1). Dose escalation and de-escalation will be guided by the BOIN design. Dose finding will continue until the pre-specified sample size of 15 is reached or stop the trial if the number of participants treated at the current dose reaches 12 and the decision is to stay at the current dose.
  Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1680mg on Day 1 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the treating investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status (e.g., symptomatic deterioration such as pain secondary to disease).
  Interventions: Drug: Iadademstat; Drug: Atezolizumab; Radiation: SBRT

INTERVENTIONS:
Drug: Iadademstat — Iadademstat is administered orally (PO) on an empty stomach (two hours after eating or one hour prior to food ingestion). After drinking the entire solution, the participant will be asked to refill the bottle with water and drink it again. Then they will drink another glass of water to wash their mouth and esophagus. Time of administration of the drug should be the same every day, preferentially in the mornings, and the time should be registered using the Dosing Instructions and Participant Drug Diary. If a dose is missed, the dose should be administered as soon as possible within 24 hours of the missed dose time. If more than 24 hours have passed, or a dose is vomited, the participant should call their medical team for instructions.
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1680mg on Day 1 (+/-3 days) of each 28-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the treating investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Administration of atezolizumab will be performed in a monitored setting where there is immediate access to trained personnel and adequate equipment and medicine to manage potentially serious reactions.
Radiation: SBRT — The first fraction of SBRT should be delivered after the initiation of iadademstat and atezolizumab, ideally between Cycle 1, Day 8, and Cycle 1, Day 15. Initiation of SBRT may be delayed up to 14 days beyond Cycle 1, Day 15 if iadademstat dose adjustment is required for toxicity

SUMMARY:
This is a phase 1b dose escalation, open-label, non-randomized study of participants with residual, progressive or recurrent ES-SCLC who previously received platinum-based chemotherapy with or without immune checkpoint inhibitor therapy; participants who have achieved only stable disease at the completion of initial platinum-based treatment are eligible for enrollment.

DETAILED DESCRIPTION:
This is a phase 1b dose escalation, open-label, non-randomized study of participants with residual, progressive or recurrent ES-SCLC who previously received platinum-based chemotherapy with or without immune checkpoint inhibitor therapy; participants who have achieved only stable disease at the completion of initial platinum-based treatment are eligible for enrollment. The primary objective is evaluating the safety, tolerability and efficacy of iadademstat combined with atezolizumab and SBRT followed by atezolizumab and iadademstat maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Ability to comply with protocol, in the treating investigator's judgment.
3. Age 18 years or older.
4. Participant must have a body weight of at least 50 Kg.
5. Histologically documented ES-SCLC previously treated with at least one regimen, including a platinum containing chemotherapy regimen, with progression of disease on or after their most recent therapy or achieving only SD after completion of one line of a platinum containing chemotherapy-based regimen.

   a. Participants previously diagnosed with limited stage SCLC treated with concurrent chemoradiation with a platinum doublet now diagnosed with recurrent extensive disease in the relapsed setting are eligible.
6. Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, antiPD-1, and anti-PD-L1 therapeutic antibodies is allowed.
7. ECOG performance status of 0 to 2.
8. At least one identified tumor lesion to be treated with SBRT.
9. At least one additional tumor lesion, separate from the site of SBRT, preferably outside of the 5Gy isodose line, amenable to incisional, excisional, core or forceps (transbronchial) biopsy. Participants must be willing to undergo tumor biopsies before starting trial therapy and 2 weeks (+/- 1 week) after the completion of SBRT.

   1. If the initial biopsy is excisional, the excised tumor cannot be counted as a biopsy target lesion and there must be another lesion amenable to incisional, excisional, core or forceps biopsy. In this scenario, the second biopsy can only be excisional if the lesion to be excised is not a target lesion.
   2. Cytology tumor specimens (e.g., from fine-needle biopsies, or drainage of pleural/ pericardial or ascites fluid) are not acceptable. Biopsies of bone lesions that do not have a soft tissue component are also not acceptable (i.e., decalcified tumor samples are not acceptable). Non-lymph node sites will be biopsied preferentially.
   3. If enrolled with stable, but not progressive, disease at the completion of first line platinum-based therapy regimen, participants may undergo biopsy of the same site that is to be irradiated. If a separate site is identified for biopsy, it should be preferentially biopsied over the site that is to be irradiated.
10. Participants must agree to submit blood samples for exploratory biomarker research at the times identified in the study calendar.
11. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can be counted as target lesions if clearly progressing after radiation.
12. Participants may have asymptomatic CNS metastases or treated CNS metastases if they are not currently receiving corticosteroids equal to or greater than prednisone 10 mg daily or equivalent for seven days prior to the first dose of study drug. Participants should have completed stereotactic radiation at least 7 days or whole brain radiation at least 2 weeks prior to Cycle 1, Day 1.

    1. Participants with new asymptomatic CNS metastases detected on their screening scan will undergo repeat CNS imaging at four weeks to ensure safety.
    2. Participants must have no history of intracranial hemorrhage or spinal cord hemorrhage from CNS disease.
    3. Metastases are limited to the cerebellum and supratentorial region (i.e. no metastases to the midbrain, pons, medulla or spinal cord).
13. Prior palliative radiotherapy must have been completed at least 1 week before the first dose of the study drug.
14. Anticonvulsants are allowed.
15. Participants must adhere to the following reproductive and contraceptive requirements while on study treatment and for at least five months after the last dose of the study drugs.

Exclusion Criteria:

1. History of leptomeningeal disease.
2. Untreated symptomatic CNS metastases. Participants with asymptomatic CNS metastases are eligible. Participant with treated symptomatic brain metastases is eligible provided they meet all of the following criteria:

   1. Completed stereotactic radiosurgery at least seven days prior to Cycle 1, Day 1 or completed whole brain radiation at least two weeks prior to Cycle 1, Day 1.
   2. No evidence of interim progression between the completion of CNS-directed therapy and the start of trial therapy.
   3. Ongoing steroid requirement of <10 mg of prednisone per day (or equivalent) as therapy for CNS disease; anticonvulsants are allowed.
   4. The participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
3. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for more than or equal to 1 week prior to enrollment.
4. Uncontrolled tumor-related pain.
5. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Participants should be recovered from the effects of radiation. There is no required minimum recovery period.
6. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
7. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

   a. Participants with indwelling catheters (e.g., PleurX) are allowed.
8. Uncontrolled or symptomatic hypercalcemia (ionized calcium greater than 1.5 mmol/L, calcium greater than 12 mg/dL or corrected serum calcium greater than ULN)
9. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 1. Preexisting Autoimmune Diseases and Immune Deficiencies for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

   1. Participants with a history of autoimmune related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   2. Participants with controlled type 1 diabetes mellitus and are on an insulin regimen will be eligible for the study.
   3. Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) are eligible for the study provided all of the following conditions are met:

   i. Rash must cover less than 10% of body surface area. ii. The disease is well controlled at baseline and requires only low-potency topical corticosteroids.

   iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
10. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

    a. History of radiation pneumonitis in the prior radiation field (fibrosis) is permitted.
11. Active tuberculosis.
12. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within three months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.

    a. Unstable angina, symptomatic or otherwise uncontrolled arrhythmia (does not include stable, alone atrial fibrillation), QTcF > 500 ms based on screening electrocardiogram (ECG), myocardial infarction ≤ 3 months prior to first study treatment, cerebrovascular accidents ≤ 3 months before study treatment start. Participant has congestive heart failure New York Heart Association (NYHA) class 2, 3 or 4 or participants with a history of congestive heart failure NYHA class 2, 3 or 4 in the past, unless a screening echocardiogram performed within one month prior to study entry demonstrates a left ventricular ejection fraction that is ≥ 45%.
13. Major surgical procedure, other than for diagnosis, within four weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
14. History of malignancy within one year prior to screening (other than SCLC), with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate greater than 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
15. Severe infection within four weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection or bacteremia.

    a. Participant has evidence of active uncontrolled viral, bacterial, or systemic fungal infection. Participants with active infection are permitted to enroll provided that the infection is clearly under control (i.e., no signs of severe systemic inflammatory response that makes participant clinically unstable in the opinion of the treating investigator, and participant is hemodynamically stable, with sustained body temperature under 38° Celsius for 48-72 hours before starting study treatment and does not need oxygen supplementation or pressors to maintain blood pressure). Participants with uncontrolled infection shall not be enrolled until the infection is treated and brought under control, as defined above.
16. Treatment with therapeutic oral or IV antibiotics within two weeks prior to initiation of study treatment.

    a. Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
17. Prior allogeneic stem cell or solid organ transplantation.
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications.
19. Treatment with a live, attenuated vaccine within four weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab or iadademstat treatment or within five months after the final dose of atezolizumab or one month after the final dose of iadademstat.
20. Current treatment with anti-viral therapy for HBV.
21. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
22. Any approved systemic anti-cancer treatment within three weeks prior to initiation of study treatment.
23. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2, IL-2) within four weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment.
24. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antiTNFagents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    1. Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after sponsor-investigator confirmation has been obtained.
    2. Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
25. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
26. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
27. Known allergy or hypersensitivity to any component of the iadademstat formulation.
28. Malabsorption syndrome or other conditions that would interfere with enteral absorption.
29. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within five months after the final dose of study treatment.
30. Known infection with HIV, HBV or HCV. Participants with prior exposure to hepatitis virus, but no evidence of active or chronic infection, may be eligible.
31. Evidence of end-organ damage as defined by the following laboratory results obtained within 14 days prior to the first study treatment:

    1. ANC <1,500 cells/µL (without granulocyte colony stimulating factor support within 14 days prior to Cycle 1, Day 1).
    2. Platelet count <100,000/µL (without transfusion within 14 days prior to Cycle 1, Day 1).
    3. Lymphocyte count < 0.75 x10^9/L.
    4. Hemoglobin <9.0 g/dL (Participants may be transfused to meet this criterion).
    5. AST, ALT, and ALP >2.5 x ULN, with the following exceptions: Participants with documented liver metastases: AST and/or ALT >5 x ULN. Participants with documented liver or bone metastases: ALP >5 x ULN.
    6. Serum bilirubin >1.5 x ULN (Participants with known Gilbert disease who have serum bilirubin level <3 x ULN may be enrolled).
    7. CrCl < 40mL/min (Cockcroft-Gault formula).
32. INR and aPTT >1.5 x ULN.

    a. This applies only to participants who are not receiving therapeutic anticoagulation; participants receiving therapeutic anticoagulation are allowed.
33. Participants with uncontrolled hypertension (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle1 Day 1 is allowed.
34. Participants receiving antidepressants reported to have KDM1A/LSD1 inhibitory activity: Tranylcypromine or Phenelzine.
35. Participants who have not recovered from grade ≥2 AEs due to prior anti-cancer therapy with the exception of alopecia, and vitiligo.
36. Participants with grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor-investigator.
37. Participants with history of clinically significant bleeding, specifically any history of intracranial hemorrhage / hemorrhagic cardiovascular accident (CVA), or participants with gastrointestinal bleeding within the 3 months prior to study entry.
38. Participants with uncontrolled disseminated intravascular coagulation.
39. Participants who refuse or are unable to potentially receive blood products.
40. Participants should be carefully questioned regarding their history of acquired or congenital immune deficiencies or autoimmune disease. Participants with any history of immune deficiencies or autoimmune disease listed in the table below are excluded from participating in the study. Possible exceptions to this exclusion could be participants with a medical history of such entities as atopic disease or childhood arthralgias where the clinical suspicion of autoimmune disease is low. Participants with a history of autoimmune related hypothyroidism on thyroid replacement hormone may be eligible for this study. In addition, transient autoimmune manifestations of an acute infectious disease that resolved upon treatment of the infectious agent are not excluded (e.g., acute Lyme arthritis). Contact the sponsor-investigator regarding any uncertainty over autoimmune exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Dose-Limiting Toxicities (DLTs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The number of participants experiencing dose-limiting toxicities (DLTs) during the study period will be recorded, providing a measure of how frequently DLTs occur when iadademstat is combined with atezolizumab and SBRT.
Rate of Dose-Limiting Toxicities (DLTs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The proportion of participants experiencing dose-limiting toxicities (DLTs), expressed as a percentage of the total participants, will be calculated. This measure aims to quantify the incidence rate of DLTs in the study population.
Grade of Dose-Limiting Toxicities (DLTs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The severity of dose-limiting toxicities (DLTs) will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. This measure will help assess the clinical significance and impact of DLTs experienced by the participants.
Frequency of Adverse Events (AEs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The number of participants experiencing adverse events (AEs) of any kind, regardless of causality, during the study period will be recorded. This outcome measure will provide insight into the overall safety profile of the combination treatment.
Rate of Adverse Events (AEs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The proportion of participants experiencing adverse events (AEs), expressed as a percentage of the total participants, will be calculated. This measure aims to quantify the incidence rate of AEs in patients treated with iadademstat combined with atezolizumab and SBRT.
Grade of Adverse Events (AEs) in patients treated with iadademstat combined with atezolizumab and SBRT | 35 days post the first dose of study drug on Cycle 1 Day 1, each cycle is 28 days long
  The severity of adverse events (AEs) will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. This measure will help assess the clinical significance and impact of AEs experienced by the participants.

SECONDARY OUTCOMES:
Disease control rate in patients treated with iadademstat combined with atezolizumab and SBRT | Measured at Cycle 2 Day 22, day 1 of subsequent cycles; where each cycle is 28 days long. Also at the survival follow up visit, which will occur 30 days post end of treatment
  Defined as the proportion of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) for a minimum duration based on RECIST v1.1 criteria (or the specific criteria used). This measure will assess the efficacy of iadademstat in combination with atezolizumab and SBRT in controlling the disease.
Objective response rate in patients treated with iadademstat combined with atezolizumab and SBRT | Measured at Cycle 2 Day 22, day 1 subsequent cycles; where each cycle is 28 days long. Also at the survival follow up visit, which will occur 30 days post end of treatment
  Defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) based on RECIST v1.1 criteria. Tumor assessments will be conducted regularly during the study to determine the ORR for patients treated with the combination of iadademstat, atezolizumab, and SBRT.
Duration of response in patients treated with iadademstat combined with atezolizumab and SBRT | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to four years
  The time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1
Progression free survival in patients treated with iadademstat combined with atezolizumab and SBRT | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to four years
  This measure will evaluate the length of time during and after treatment that the patient lives without disease progression when treated with iadademstat, atezolizumab, and SBRT.
Overall Survival (OS) in patients treated with iadademstat combined with atezolizumab and SBRT | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to four years
  Measured from the date of treatment initiation until the date of death from any cause. This outcome measure will help determine the overall longevity of patients following treatment with the combination of iadademstat, atezolizumab, and SBRT.
Local Control of Irradiated Target Lesion in patients treated with iadademstat combined with atezolizumab and SBRT | At Cycle 2 Day 22 then on Day 1 of subsequent cycles, where each cycle is 28 days. Finally, at the survival follow up visit, which will occur 30 days post end of treatment
  To assess the local control of the irradiated target lesion when stereotactic body radiotherapy (SBRT) is administered in combination with iadademstat and atezolizumab. This determination will be made by the treating investigator according to RECIST v1.1 criteria applied specifically to the irradiated lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Annie Chiang, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No